CLINICAL TRIAL: NCT01349894
Title: Post-Market Clinical Evaluation of the Spiracur SNaP™ Wound Care System for Treatment of Skin Cancer Excision Sites and Split Thickness Skin Grafts
Brief Title: SNaP Wound Care System Over Skin Cancer Excision Sites and Split Thickness Skin Grafts (STSGs)
Status: Withdrawn | Type: Observational
Why Stopped: The study was terminated by Spiracur (original sponsor). Efforts were made to contact the PI/study team members, but were unsuccessful.
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: 011111
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Split Thickness Skin Graft; Skin Cancer Excision Site; Skin Graft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SNaP® Wound Care System
  Interventions: Device: SNaP® Wound Care System

INTERVENTIONS:
Device: SNaP® Wound Care System — Wound dressing applications using customized system. Dressing applications changes per manufacturer recommendation.

SUMMARY:
The purpose of this study is to evaluate the efficacy of the Spiracur SNaP® Wound Care System for the treatment of skin cancer excision sites and split thickness skin grafts (STSG). The secondary purpose will be to compare the prospective patients to retrospectively treated skin cancer excision sites and STSGs to further evaluate efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Skin cancer excision site and/or STSG as the source of the wound on any part of the body including head and neck, torso, and extremities. Any other type of skin graft will also be eligible for inclusion into the study.
* Wound < 16 cm in greatest diameter
* Subject ≥ 18 years of age
* Female subjects of child-bearing potential must be willing to take a urine pregnancy test prior to starting study
* Subject is willing and able to sign informed consent

Exclusion Criteria:

* Wound-related cellulitis
* Wound located in an area not amenable to forming an air-tight seal
* Subject has untreated osteomyelitis
* Subject is allergic to wound care products
* Wound has exposed blood vessels not suitable for negative pressure therapy
* Subject is actively participating in other clinical trials that conflict with current study
* Subject has fistulas
* Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from existing investigator patient population.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Wound Closure | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francis Papay, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Dermatology and Plastic Surgery Institute, Cleveland Clinic, Cleveland, Ohio, United States